CLINICAL TRIAL: NCT01660256
Title: Confirmatory Study of OPC-12759 Ophthalmic Solution in Patients With Dry Eye
Brief Title: Confirmatory Study of OPC-12759 Ophthalmic Solution
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 037E-11-003; JapicCTI-121920 (Other: JapicCTI)
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Results first posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — rebamipide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- OPC-12759 ophthalmic solution (Experimental): OPC-12759 ophthalmic solution
  Interventions: Drug: OPC-12759
- Placebo (Placebo Comparator): OPC-12759 ophthalmic solution 0%
  Interventions: Drug: Placebo
- OPC-12759 ophthalmic suspension (Active Comparator): OPC-12759 ophthalmic suspension
  Interventions: Drug: OPC-12759

INTERVENTIONS:
Drug: OPC-12759 — Instillation, 4 times/day for 4 weeks
  Other Names: rebamipide
  Arms: OPC-12759 ophthalmic solution; OPC-12759 ophthalmic suspension
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to verify whether OPC-12759 ophthalmic solution is effective compared with placebo in dry eye patients. OPC-12759 ophthalmic suspension will be used as a reference drug.

ELIGIBILITY:
Inclusion Criteria:

1. Out patient
2. Subjective complaint of dry eye that has been present for minimum 20 months
3. Ocular discomfort severity is moderate to severe
4. Corneal - conjunctival damage is moderate to severe
5. Unanesthetized Schirmer's test score of 5mm/5minutes or less
6. Best corrected visual acuity of 0.2 or better in both eyes

Exclusion Criteria:

1. Presence of anterior segment disease or disorder other than that associated with dry eye
2. Ocular hypertension patient or glaucoma patient with ophthalmic solution
3. Anticipated use of any topically-instilled ocular medications or patients who cannot discontinue the use during the study
4. Anticipated use of contact lens during the study
5. Patient with punctal plug
6. Any history of ocular surgery within 12 months
7. Female patients who are pregnant,possibly pregnant or breast feeding
8. Known hypersensitivity to any component of the study drug or procedural medications
9. Receipt of any investigational product within 4 months.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2012-08; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eiji Murakami, Study Director — Director of Division Dermatilogicals and Ophtalmolgicals, Otsuka Pharmaceutical Co., Ltd.
Locations (4):
- Japan (4):
  - Kansai Region, Kansai Region
  - Kanto region, Kanto Region
  - Kyushu region, Kyushu Region
  - Tokai region, Tokai Region

RESULTS

PARTICIPANT FLOW:
Groups:
- OPC-12759 Solution: One drop of 2% OPC-12759 ophthalmic solution was instilled into each eye 4 times a day for 4 weeks.
- Placebo: One drop of 0% OPC-12759 ophthalmic solution was instilled into each eye 4 times a day for 4 weeks.
- OPC-12759 Suspension: One drop of 2% OPC-12759 ophthalmic suspension was instilled into each eye 4 times a day for 4 weeks.
Period: Overall Study
Arm/Group | OPC-12759 Solution | Placebo | OPC-12759 Suspension
Started | 84 | 83 | 42
Completed | 79 | 83 | 38
Not Completed | 5 | 0 | 4
Not completed — Adverse Event | 4 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OPC-12759 Solution | Placebo | OPC-12759 Suspension | Total
Number analyzed (Participants) | 84 | 83 | 42 | 209
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (18.6) | 56.5 (16.6) | 54.2 (16.8) | 56.5 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 67 | 35 | 176
  Male | 10 | 16 | 7 | 33
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 84 | 83 | 42 | 209

OUTCOME MEASURES:

1. Primary Outcome: Change in Fluorescein Corneal Staining (FCS) Score From Baseline
Description: FCS indicates the damage to the corneal epithelium. Per the National Eye Institute/Industry Workshop report, the cornea was divided into 5 fractions, each of which was given a staining score from 0 to 3, and the total score was calculated (0-15). 0 is better.
  Changes of the FCS score from baseline to the last dose (last observation carried forward [LOCF]) were compared between 2% OPC-12759 ophthalmic solution and placebo by the t-test.
Time Frame: Baseline, Week 4
Population: Full analysis set consisted of all subjects who had received the investigational product at least once after randomized assignment to a treatment group.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | OPC-12759 Solution | Placebo | OPC-12759 Suspension
Number analyzed (Participants) | 84 | 83 | 42
score on a scale | -3.3 (0.2) | -2.0 (0.3) | -2.9 (0.3)
Statistical Analysis 1: Comparison: OPC-12759 Solution vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -1.3

2. Secondary Outcome: Change in Lissamine Green Conjunctival Staining (LGCS) Score From Baseline
Description: LGCS indicates the damage to the conjunctival epithelium. Per the National Eye Institute/Industry Workshop report, the conjunctiva was divided into 6 fractions, each of which was given a staining score from 0 to 3, and the total score was calculated (0-18). 0 is better.
  The scores and change from baseline at each examination (including LOCF) were compared between 2% OPC-12759 ophthalmic solution and placebo ophthalmic solution.
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | OPC-12759 Solution | Placebo | OPC-12759 Suspension
Number analyzed (Participants) | 84 | 83 | 42
score on a scale | -3.2 (0.3) | -1.7 (0.3) | -3.1 (0.4)
Statistical Analysis 1: Comparison: OPC-12759 Solution vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -1.5

ADVERSE EVENTS:
Time Frame: Treatment period (4 weeks)
Description: Only adverse events that occurred after the start of study treatment were evaluated.
  Safety analysis set consisted of all subjects who had received the investigational product at least once.
Arm/Group | OPC-12759 Solution | Placebo | OPC-12759 Suspension
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/83 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/83 | 0/42
Other Adverse Events (participants affected / at risk) | 23/84 | 11/83 | 11/42
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-12759 Solution (N=84) | Placebo (N=83) | OPC-12759 Suspension (N=42)
Abnormal sensation in eye (Eye disorders) | 1 | 0 | 1
Eye irritation (Eye disorders) | 0 | 0 | 1
Ocular discomfort (Eye disorders) | 1 | 0 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Periproctitis (Gastrointestinal disorders) | 0 | 1 | 0
Adenoviral conjunctivitis (Infections and infestations) | 0 | 0 | 1
Hordeolum (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 5 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
Glucose urine present (Investigations) | 1 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0
Protein urine present (Investigations) | 1 | 0 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 13 | 1 | 5
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No